CLINICAL TRIAL: NCT05694806
Title: Clinical Impact of Thoracic Scanographic Characteristics of Hematologic Malignancy Patients with Mediastinal Mass Syndrome Admitted to the Intensive Care Unit
Brief Title: Clinical Impact of Thoracic Scanographic Characteristics of Hematologic Malignancy Patients
Acronym: MED-HEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0237
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Mediastinal Diseases
Keywords: Mediastinal mass syndrome
MeSH Terms: conditions — Mediastinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with symptomatic Mediastinal mass syndrome: patients with symptomatic Mediastinal mass syndrome at diagnosis or at relapse of a patient with haematological malignancy admitted to the Intensive Care unit
  Interventions: Other: analysis of thoracic scans

INTERVENTIONS:
Other: analysis of thoracic scans — analysis of thoracic scans realised in standard care

SUMMARY:
The mediastinum can be the site of benign or malignant tumors, including 10 to 20% of hematological malignancies.

Mediastinal mass syndrome (MMS) includes symptoms due to irritation, invasion or compression of the organs of the mediastinum. This syndrome includes respiratory manifestations that may be secondary to compression of the tracheobronchial tree, venous vascular manifestations with the superior vena cava syndrome or arterial manifestations, cardiac manifestations, digestive or nervous manifestations.

The management of a mediastinal syndrome is a diagnostic and therapeutic emergency requiring the collaboration of several disciplines in order to achieve the most effective but least deleterious way possible to diagnostic imaging, etiological biopsy, and the possible implementation of life-saving symptomatic measures before the initiation of etiological treatment.

Diagnostic thoracic imaging relies primarily on thoracic computed tomography (CT) to determine the size and nature of the mediastinal mass, the presence and extent of tracheobronchial or great vessel compression, the presence of pleural and/or pericardial effusion, pulmonary embolism, parenchymal lesions, and possibly subdiaphragmatic lesions.

However, the potential severity of MMS is often under-diagnosed in adult patients, particularly in the context of hematologic malignancy. Indeed, we have very little literature on the initial management of these patients at risk.

The present study propose to conduct the first multicenter study to analyze the characteristics (clinical, scanographic, echocardiographic, hematological and resuscitation) of the initial management of patients with symptomatic MMS at diagnosis or at relapse of a patient with MH admitted to the Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancy at diagnosis or relapse
* Symptomatic mediastinal mass syndrome
* Admission to the ICU, Continuous Medical Surveillance (CMS) or Intensive Care (IC) for symptomatology related to MMS
* Chest CT (after maximum 48 hours of corticosteroid therapy (1mg/kg/ Prednisone equivalent), maximum 15 days before and 5 days after admission to ICU)
* Maximum administration of corticosteroid therapy 48 hours before admission to the ICU (maximum 1mg/kg/ Prednisone equivalent)
* No prior pleural or pericardial drainage
* Study period: 01/01/2014 - 31/12/2021 (8 years)

Exclusion Criteria:

* No diagnosis of hematologic malignancy
* Diagnosis of solid benign or malignant tumor
* No mediastinal mass syndrome
* No admission to ICU/CMS
* No chest CT scan meeting inclusion criteria
* Administration of corticosteroids for more than 48 hours prior to admission to the ICU and/or prior to chest CT
* Lack of social security affiliation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with eligibility criteria hospitalised during the study period 01/01/2014 - 31/12/2021
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To identify prognostic thoracic scan factors of severe mediastinal mass syndrome | 1 week
  To identify prognostic thoracic scan factors of severe mediastinal mass syndrome defined by the occurrence of severe respiratory, hemodynamics and/or neurological failures.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Picard, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Muriel Picard, Toulouse, France

IPD SHARING:
Plan to Share IPD: No